CLINICAL TRIAL: NCT06257693
Title: A Phase 1 Study to Establish the Feasibility of Enolen (tm) for the Local Delivery of Enzalutamide in Patients With Prostate Cancer
Brief Title: Enzalutamide Implants (Enolen) in Patients With Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alessa Therapeutics Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP-001; ZIABC011081 (NIH)
Record Dates: First submitted 2023-12-14; First posted 2024-02-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enolen (tm) (Experimental): Enolen (tm) implants containing enzalutamide
  Interventions: Drug: enzalutamide

INTERVENTIONS:
Drug: enzalutamide — Localized single delivery of the Enolen implant (polymer + enzalutamide) with planned radical prostatectomy
  Other Names: Radical prostatectomy

SUMMARY:
The study is to assess whether the Enolen is safe and delivers anti-androgen medication locally in patients that are planning for radical prostatectomy.

DETAILED DESCRIPTION:
This study is a multi-center, open-label feasibility study. Up to 56 participants planning for radical prostatectomy will be recruited to assess the safety and patient tolerance of Enolen for the localized delivery of enzalutamide into the prostate.

At baseline, patients will undergo multiparametric MRI of the prostate. Study participants will have placement of the drug eluting Enolen implants followed by a standard of care prostatectomy 6-12 weeks or 4-12 months post-implant procedure.

Twenty participants in Cohort A receive up to 16 implants and have a prostatectomy planned between weeks 6 and 12 post-implant procedure.

Twenty-four participants in Cohort B are randomized to 8 or 16 implants and have a prostatectomy planned between weeks 6 and 12 post-implant procedure.

Twelve participants in Cohort C receive 16 implants and have a prostatectomy planned between months 4 and 12 post-implant procedure. If the participant is unwilling to undergo the prostatectomy by 12 months, they must agree to close monitoring with imaging by MRI every three months and biopsies, as indicated, for up to 24 months post-implant procedure.

Study participants are followed for 2-6 weeks post-prostatectomy.

Participants will be followed for an additional 6-12 weeks post surgery. Clinical labs and correlative sample collection and patient quality of life questionnaires will be administered at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 21 years old
2. Histologically confirmed adenocarcinoma of the prostate
3. Study participant qualified and planning for radical prostatectomy
4. At least 1 prostate lesion measurable by MRI greater or equal to 0.5 cm
5. Cohort A and Cohort B: Gleason score 3+4 or higher Cohort C: Gleason score 3+3 with high risk features or 3+4
6. Study participant must be willing to undergo post-treatment imaging by MRI
7. Participants must be able to understand and sign the informed consent form
8. ECOG performance status 0 or 1
9. Adequate organ function, including absolute neutrophil count (ANC) ≥1000 cells/μL, hemoglobin ≥9 g/dL, platelets ≥100,000 cells/μL, estimated creatinine clearance ≥50 mL/min, bilirubin <1.5x ULN (< 3x ULN for documented Gilbert's syndrome)
10. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and Alkaline phosphatase <2.5x ULN
11. The effects of Enolen on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, men must agree to use a highly effective form of contraception or abstinence at the time of study entry and continuing through three months after radical prostatectomy/implant removal. Highly effective forms of contraception include:

Vasectomy Condom with spermicide

Partner use of one of the following methods:

Postmenopausal >1 year or age >55y Bilateral tubal ligation Intrauterine devices (IUDs) Hormonal implants (Implanon, Nexplanon, etc.) Combination oral contraceptives Progestin-only injections (Depo-Provera) Hormonal patches Vaginal Ring Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, the treating physician should be informed immediately.

Exclusion Criteria:

1. Prior radiotherapy or surgery for prostate cancer
2. Ongoing hormonal therapy for prostate cancer or hormone therapy <3 months prior to the start of treatment
3. Prior prostate procedures such as transurethral resection of the prostate, transurethral microwave thermotherapy of the prostate, high-intensity focused ultrasound or minimally invasive Benign Prostate Hyperplasia (BPH) procedure
4. Study participant unwilling or unable to undergo MRI, including participants with contra-indications to MRI, such as cardiac pacemakers, non-compatible intracranial vascular clips, etc.
5. Metallic hip implant or any other metallic implant or device that distorts the quality of prostatic MR images.
6. Study participants who, because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent.
7. Presence of any metastatic disease.
8. No evidence of extracapsular extension of disease.
9. Study participants, who in the opinion of the treating clinician, would be at increased risk of refractory urinary retention due to a transperineal procedure such as the Enolen implant.
10. History of prostate infection within 2 years.
11. No intercurrent medical condition or circumstances that would preclude prostatectomy.
12. History of bleeding diathesis or currently on anti-coagulation therapy that cannot be safely discontinued for implant procedure.
13. Any condition that, in the opinion of the Principal Investigator, which would impair the participant's ability to comply with study procedures and undergo prostatectomy.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
To assess the adverse events associated with the Enolen implant | up to 12 months
  Using Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v.5.0).
Measurement of Pharmacokinetics Profile | up to 12 months
  Enzalutamide plasma (ng/ml) and tissue levels (ng/gm)

SECONDARY OUTCOMES:
MRI changes | up to 12 months post Enolen implantation
  Prostate and tumor volume changes (mm3)
Changes in Prostate-specific antigen (PSA) | 6 to 12 weeks post radical prostatectomy
  Measurements of the amount of PSA in the blood (ng/ml) at baseline through 6-12 weeks post radical prostatectomy
Changes in Testosterone | 6 to 12 weeks post Enolen implantation
  Measurements of testosterone levels in the blood (ng/dl) from baseline to radical prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pinto, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (7):
- United States (7):
  - Northwestern University, Chicago, Illinois
  - Mary Bird Cancer Center, Metairie, Louisiana
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - VA Portland Health Care System, Portland, Oregon
  - Atlantic Urology Specialists, Myrtle Beach, South Carolina
  - Virginia Commonwealth University, Richmond, Virginia
  - Aurora Urology, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Alessa Therapeutics will allow NCI to share data, including genomic data, on this project.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data is shared after the completion of the study.
Access Criteria: Data will be provided by the sponsor/Alessa Therapeutics to the NIH for sharing per the NIH Data Managment and Sharing Policy